CLINICAL TRIAL: NCT05297812
Title: Alpha-1 Antitrypsin Disease Cohort: Longitudinal Biomarker Study of Disease - Alpha-1 Biomarker Research Consortium (A1BC)
Brief Title: Alpha-1 Antitrypsin Disease Cohort: Longitudinal Biomarker Study of Disease
Acronym: A1BC
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Alpha-1 Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeanine D'Armiento, Associate Professor of Medicine (in Anesthesiology), Columbia University
Other Study IDs: AAAS8713; 1UG3HL152323 (NIH)
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alpha 1-Antitrypsin Deficiency; Genetic Disease
Keywords: Alpha-1; Biomarker; PiZZ
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Blood samples will be collected for analysis in the ongoing clinical trial as well as for banking to for a bio-repository for future AATD studies. Participants will have the option to agree/not agree to partake in the optional bio-repository.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate to Advanced Emphysema: Patients with moderate or advanced Emphysema as measured by baseline inspiratory PERC-15 below the study median
- Minimal Emphysema: Patients with minimal emphysema as measured by baseline inspiratory PERC-15 above the study median

SUMMARY:
Alpha-1 Anti-trypsin Deficiency (AATD) is a genetic disease with lung and liver disease presentations. The purpose of this study is to examine the density of the lung as measured by chest computed tomography (CT) and determine if existing emphysema predicts changes in the rate of subsequent emphysema or changes in CT, serum or plasma biomarkers of interest. The overarching goal is to develop biomarkers that can be used in interventional trials since lung function changes do not typically inform disease progression in AATD.

DETAILED DESCRIPTION:
Progression of lung disease in patients with Alpha-1 Anti-trypsin deficiency is variable and while some patients may have stable lung function over many years, some progress and deteriorate rapidly. Currently there are no predictors that would help identify patient at risk of rapid deterioration. The aim of this study is to identify markers and features in CT imaging that may allow identification of these patients early before deterioration. To achieve this, the study will follow a cohort of patients with confirmed Alpha-1 Anti-trypsin deficiency and lung disease and measure a number of biomarkers in blood and sputum and obtain high resolution CT scans at baseline and again three years later. If the study is able to determine markers that allow the identification of patients at risk early, the investigator may be able to study early interventions in later studies and possibly find ways to avoid serious complications. Patients will be followed longitudinally to assess deterioration of lung function.

Study procedures include: Review of medical history and medication history, blood draw, complete Pulmonary Function Test (PFT), induced sputum (at some sites), completion of questionnaires and CT Chest scan. All of the mentioned procedures above will be performed on enrollment and repeated at 18 months and 36 months, with the exception of monthly Alpha- net exacerbation questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 years and older
2. Patients with known Alpha-1 Anti-trypsin deficiency (PiZZ)
3. Be an existing member of the Alpha-1 Foundation Clinical Cohort (Alpha-1 Foundation Research Registry)
4. Willingness to perform study procedures of Chest CT, blood biomarker determination, questionnaire completion, and lung function testing.

Exclusion Criteria:

1. AATD non-PiZZ status, including carriers
2. Pregnancy at the time of the screening visit
3. COPD exacerbation or other pulmonary infection within 6 weeks of baseline visit
4. Previous lung or liver transplantation or currently on the transplant list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alpha-1 Antitrypsin Deficiency genotype ZZ across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in lung density over three years | 3 years
  Change in lung density over three years determined by using the 15th percentile point of Hounsfield units in inspiratory high resolution CT scans (PERC-15)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine M D'Armiento, MD, PhD, Principal Investigator — Columbia University; Charlie Strange, MD, Study Chair — Medical University of South Carolina
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Boston University, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
This study is part of a larger research study where one of the objectives is to create a AATD de-identified, public use repository of data. This repository will be query based, and any sub-projects that stem from this will need to abide by the appropriate Human Subjects Protection, GCP guidelines (i.e., IRB protocol, local IRB approval, DUA, Release of Information) and be reviewed by the research committee including the Alpha-1 Foundation prior to release of any de-identified data.
Supporting Information: Study Protocol
Time Frame: After first 3 years of data collection and preliminary analysis
Access Criteria: De-identified data will be available via i2b2 with proper protocol and IRB regulatory documentation